CLINICAL TRIAL: NCT06963892
Title: Examining the Effect of Neuromuscular Exercises on Movement Control in Hip & Knee Osteoarthritis: A Randomised Proof of Concept and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71072.A1; 306886 (Other: The Integrated Research Application System (IRAS))
Record Dates: First submitted 2023-08-24; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis; Hip; Knee OA; Motor Control
Keywords: Hip and Knee Osteoarthritis; Movement Control; Movement Screening Tools; Neuromuscular Exercise; Feasibility Study; Proof of Concept
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuromuscular Exercise Intervention (Experimental): Participants attended six supervised group exercise sessions over six weeks. Each session (~60 min) included structured neuromuscular exercises focusing on joint stability, functional movement retraining, balance, proprioception, and muscle strengthening, following principles from the Good Life with osteoArthritis in Denmark (GLA:D®) programme. Exercises were progressed based on individual capability and pain tolerance.
  Interventions: Behavioral: Neuromuscular Exercise Programme (GLA:D®-based
- Usual Physiotherapy Care (Active Comparator): Participants received usual care provided by NHS physiotherapy outpatient services. This involved standard joint mobility exercises, strengthening activities, general advice, and education typically offered to patients with hip or knee osteoarthritis, without specific emphasis on structured neuromuscular control training.
  Interventions: Behavioral: Usual Physiotherapy Care (NHS Standard)

INTERVENTIONS:
Behavioral: Neuromuscular Exercise Programme (GLA:D®-based — Participants underwent supervised neuromuscular exercise sessions based on the Good Life with osteoArthritis in Denmark (GLA:D®) programme. Exercises targeted dynamic joint stability, balance, proprioception, functional movements, and muscle strengthening. Sessions were held once weekly, lasting approximately 60 minutes each, over six consecutive weeks. The intervention was tailored progressively to each participant's capabilities, symptoms, and pain tolerance.
  Other Names: Neuromuscular training; sensorimotor exercise
  Arms: Neuromuscular Exercise Intervention
Behavioral: Usual Physiotherapy Care (NHS Standard) — Participants received standard NHS physiotherapy care for hip or knee osteoarthritis. This included routine joint mobility exercises, strengthening activities, general education, and advice. Sessions were delivered in outpatient clinics following standard practice without specific emphasis on neuromuscular control training. Frequency and duration-matched usual clinical care.
  Other Names: Routine physiotherapy, Standard OA physiotherapy
  Arms: Usual Physiotherapy Care

SUMMARY:
This completed study evaluated the effects of a six-week neuromuscular exercise programme on movement control in individuals with hip and/or knee osteoarthritis (OA). The trial also assessed the feasibility of conducting a future definitive randomised controlled trial.

A total of 90 participants with symptomatic hip or knee OA were recruited from NHS outpatient physiotherapy clinics and cluster-randomised to either an intervention group or a control group. The intervention group received a structured neuromuscular exercise programme based on the GLA:D® approach, delivered once weekly for six weeks. The control group received usual care, including general physiotherapy advice and standard exercises.

The primary outcome was change in movement control, assessed using the Short Hip and Lower Limb Movement Screen (Short-HLLMS) at baseline and six weeks. Secondary outcomes included joint-specific function measured by KOOS-12 and HOOS-12 questionnaires, and pain intensity assessed using the Numeric Pain Rating Scale (NPRS). Feasibility measures included recruitment rate, participant adherence, and study retention.

The study was completed successfully and demonstrated that neuromuscular exercise may improve short-term movement control and functional outcomes in individuals with OA. Feasibility outcomes supported the acceptability of the intervention and the procedures for conducting a future large-scale trial.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic joint condition that significantly impacts mobility, function, and quality of life. Although exercise is strongly recommended in clinical guidelines for managing OA, the specific role of neuromuscular training-exercises targeting sensorimotor control, functional movement patterns, and joint stability-has not been thoroughly investigated in terms of improving movement control in this population. Previous research indicates that compromised neuromuscular control may contribute to altered biomechanics, increased joint loading, pain, and functional limitations among people with OA. However, structured neuromuscular interventions aiming explicitly at enhancing movement control remain understudied in clinical practice.

This study addressed this gap by conducting a cluster-randomised, proof-of-concept and feasibility trial designed to evaluate the effects of a structured neuromuscular exercise intervention based on principles from the Good Life with osteoArthritis in Denmark (GLA:D®) programme. This exercise programme has previously shown benefits in reducing OA symptoms and improving function, but its effect on movement control using structured assessments has yet to be explored.

Participants with clinically diagnosed symptomatic hip or knee OA were recruited from NHS physiotherapy outpatient clinics in the United Kingdom. Following recruitment, study sites were cluster-randomised to either the intervention or control group to minimise cross-group contamination. Participants at sites allocated to the intervention group underwent a supervised, structured neuromuscular exercise programme delivered by trained physiotherapists. This programme involved six supervised sessions, conducted once per week, with each session lasting approximately 60 minutes. Each session comprised a brief educational component followed by exercises focusing on dynamic joint stability, functional movement retraining, proprioception, balance, and muscle strengthening.

The neuromuscular exercises were progressively adjusted to individual abilities and pain tolerance, with careful monitoring of participants to ensure exercises were performed safely and correctly. Training intensity and exercise difficulty gradually increased throughout the intervention period, adhering closely to the established protocol from the GLA:D® programme.

Participants at control sites received standard physiotherapy care typically provided to individuals with hip or knee OA within the NHS. This standard care included general joint mobility exercises, strength training, general physiotherapy advice, and education provided during routine outpatient appointments.

To assess the impact of the neuromuscular exercise programme, the study used a novel clinical screening tool known as the Short Hip and Lower Limb Movement Screen (Short-HLLMS). This observational tool evaluates key movement patterns such as squatting and single-leg activities, providing a structured approach to identify movement impairments related to joint stability, coordination, and alignment.

Additionally, feasibility outcomes such as participant recruitment rates, retention, adherence to the intervention, and overall acceptability of the neuromuscular exercises were systematically evaluated to inform the potential for scaling up the intervention in future larger-scale trials or clinical practice implementation. Participant experiences and perceptions of the intervention were collected to understand barriers and facilitators to participation, adherence, and potential clinical translation.

The study aimed primarily to establish proof-of-concept regarding neuromuscular training's potential effectiveness in improving movement control, a crucial outcome associated with joint health and functional independence. This study also aimed to identify practical considerations essential for conducting a definitive randomised controlled trial, such as realistic recruitment timelines, dropout rates, and adherence to structured exercise programmes.

The results of this feasibility study have implications for both clinical practice and future research, providing evidence on whether a neuromuscular exercise approach can meaningfully influence movement quality in patients with hip and knee OA and inform decision-making for subsequent research phases, including larger-scale effectiveness trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 years or older.
* Clinically diagnosed symptomatic hip and/or knee osteoarthritis (unilateral or bilateral).
* Meeting the American College of Rheumatology (ACR) clinical criteria for osteoarthritis.
* Able to safely participate in neuromuscular exercises and movement screening tests.

Exclusion Criteria:

* Acute septic arthritis.
* Inflammatory arthritis (e.g., rheumatoid arthritis).
* Avascular necrosis of the hip or knee.
* Recent steroid injections (within the past 3 months).
* Knee or hip surgery within the previous 12 months.
* Significant cardiorespiratory or systemic disorders limiting exercise participation.
* Neurological conditions (e.g., stroke, Parkinson's disease, multiple sclerosis).
* Body mass index (BMI) greater than 35 kg/m².
* Severe low back pain restricting activity.
* Cognitive impairment affecting ability to follow study instructions.
* Skin conditions affecting lower limbs, preventing safe participation in exercises.
* Inability to communicate effectively in English or understand the consent information.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Change in movement control measured by the Short Hip and Lower Limb Movement Screen (Short-HLLMS) | Baseline (pre-intervention) and at 6 weeks (post-intervention)
  The Short Hip and Lower Limb Movement Screen (Short-HLLMS) was used to objectively assess participants' movement control, alignment, and joint stability. The screen evaluated three functional tasks: small knee bend, standing hip flexion, and deep squat. Lower scores indicate better movement quality and control. Assessments were performed at baseline (pre-intervention) and immediately following the six-week intervention period (post-intervention). The primary outcome measure was the change in Short-HLLMS scores from baseline to six weeks.

SECONDARY OUTCOMES:
Change in Knee-specific Function (KOOS-12) | Baseline (pre-intervention) and at 6 weeks (post-intervention)
  The Knee Injury and Osteoarthritis Outcome Score Short-form (KOOS-12) questionnaire measured patient-reported knee-specific function, pain, and quality of life. Scores range from 0 to 100, with higher scores indicating better knee function and reduced symptoms.
Change in Hip-specific Function (HOOS-12) | Baseline (pre-intervention) and at 6 weeks (post-intervention)
  The Hip Disability and Osteoarthritis Outcome Score Short-form (HOOS-12) questionnaire measured patient-reported hip-specific function, pain, and quality of life. Scores range from 0 to 100, with higher scores representing better hip function and reduced symptoms.
Change in Pain Intensity (Numeric Pain Rating Scale) | Baseline (pre-intervention) and at 6 weeks (post-intervention)
  Pain intensity was assessed using the Numeric Pain Rating Scale (NPRS), which is a valid patient-reported measure of pain severity. Scores range from 0 (no pain) to 10 (worst imaginable pain). Lower scores indicate reduced pain severity.
Feasibility of the Intervention (Recruitment and Retention Rates) | Measured continuously during recruitment and across the 6-week intervention period
  Feasibility outcomes included the percentage of eligible patients who consented to participate, adherence to the intervention (measured by attendance rates), and the dropout rate during the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Umer Umer Sheikh, MSc, Principal Investigator — University of Southampton, School of Health Sciences
Locations (1):
- Ashford & St Peters NHS Hospital, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We need to discuss this first

REFERENCES:
- [Background] Abramoff B, Caldera FE. Osteoarthritis: Pathology, diagnosis, and treatment options. Med Clin North Am. 2020;104(2):293-311. Ageberg E, Roos EM. Neuromuscular exercise as treatment of degenerative knee disease. Exerc Sport Sci Rev. 2015;43(1):14-22. Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualised goal-based NEMEX-TJR training programme. BMC Musculoskelet Disord. 2010;11(1):126. Ageberg E, Nilsdotter A, Kosek E, Roos EM. Effects of neuromuscular training (NEMEX-TJR) on function and quality of life in individuals with hip and knee osteoarthritis: A randomised controlled trial. Osteoarthritis Cartilage. 2010;18(8):971-6. Atkinson G, Nevill AM. Selected issues in the design and analysis of sport performance research. J Sports Sci. 2001;19(10):811-27. Booysen N, Wilson DA, Lewis CL, Warner MB, Gimpel M, Mottram S, et al. Assessing movement quality using the hip and lower limb movement screen: development, reliability and potential applications. J Musculoskelet Res. 2019;22(3-4):1950008. King LK, Birmingham TB, Callaghan JP, et al. Personalised neuromuscular interventions in osteoarthritis rehabilitation: A step toward precision medicine. J Orthop Res. 2023;41(5):789-804. Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D®): Evidence-based education and supervised neuromuscular exercise for patients with knee and hip osteoarthritis. BMC Musculoskelet Disord. 2017;18(1):72. Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, et al. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007;15(9):981-1000. Gandek B, Roos EM, Franklin PD, Ware JE. A 12-item short form of the Knee injury and Osteoarthritis Outcome Score (KOOS-12): tests of reliability, validity and responsiveness. Osteoarthritis Cartilage. 2019;27(5):762-70. Gandek B, Roos EM, Franklin PD, Ware JE. A 12-item short form of the Hip disability and Osteoarthritis Outcome Score (HOOS-12): tests of reliability, validity and responsiveness. Osteoarthritis Cartilage. 2019;27(5):754-61.